CLINICAL TRIAL: NCT01200602
Title: A Randomized Megestrol Acetate/Placebo Controlled Trial in Pediatric Patients With Malignancies With Weight Loss/Anorexia
Brief Title: Megestrol Acetate in Treating Weight Loss or Anorexia in Young Patients With Malignancies Who Are Undergoing Radiation Therapy and/or Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study closed due to slow accrual.
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC0896; NCI-2010-01938 (Registry Identifier: NCI-CTRP); 09-007533 (Other: Mayo Clinic IRB); MC0896 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2010-09-10; First posted 2010-09-13 (Estimated); Results first posted 2013-05-24 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Anorexia; Weight Changes
MeSH Terms: conditions — Anorexia; Body Weight Changes | interventions — Megestrol Acetate; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Patients receive oral megestrol acetate 1-2 times daily for 4 weeks.
  Interventions: Drug: megestrol acetate
- Arm B (Active Comparator): Patients have clinical observation for weight loss and gain for 4 weeks.
  Interventions: Other: clinical observation

INTERVENTIONS:
Drug: megestrol acetate — Given orally in doses of either 10 mg/kg once a day or 5 mg/kg twice a day
  Other Names: BDH 1298; Maygace; Megace; Megestil; Niagestin; Pallace
  Arms: Arm A
Other: clinical observation — No treatment is given.
  Other Names: observation
  Arms: Arm B

SUMMARY:
RATIONALE: Megestrol acetate may help improve appetite and lessen weight loss caused by cancer. PURPOSE: This clinical trial studies megestrol acetate in treating weight loss or anorexia in young patients with malignancies who are undergoing radiation therapy and/or chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:Proportion of Patients Who Maintain Weight or Experience Weight Gain.

SECONDARY OBJECTIVES:BMI Trends, Caloric Intake, Weight Maintenance Over Time, Toxicity Profile as Assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v.4.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM A: Patients receive oral megestrol acetate 1-2 times (10 mg/kg dose if once daily or 5 mg/kg dose if twice daily) daily for 4 weeks. ARM B (control): Patients are observed for weight loss and gain for 4 weeks. After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric patient with an underlying diagnosis of a malignancy (excluding hematological malignancies like leukemias and lymphomas)
* ≥5% weight loss from diagnosis of primary malignancy (must be currently on chemotherapy and/or radiation therapy or scheduled to receive cancer therapy OR ≥5% weight loss following bone marrow transplant (autologous or allogeneic blood/bone marrow) and not actively receiving corticosteroid therapy
* Negative pregnancy test done =< 7 days prior to registration for women of childbearing potential only

Exclusion Criteria:

* Receiving tube feedings or parenteral nutrition
* Evidence of ascites
* Current (within the past 28 days) or planned treatment with adrenal steroids (short-term use of dexamethasone around days of intravenous chemotherapy is allowed for protection against emesis), androgens, progestational agents, or appetite stimulants (e.g., dronabinol)
* Known mechanical obstruction of the alimentary tract, malabsorption, or intractable vomiting (> 5 episodes/week)
* History of unresectable brain tumor or cancer metastatic to the brain
* History of thromboembolic disease
* Insulin-requiring diabetes
* Congestive heart failure and/or uncontrolled hypertension
* Anticoagulation
* Previous history of thrombosis (personal and immediate family)
* Concurrent corticosteroid therapy (except as an antiemetic)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vilmarie Rodriguez, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One patient was accrued between March 2, 2011 and January 10, 2012. Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Sex: Female, Male [Count of Participants; unit: Participants] — Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Region of Enrollment [Number; unit: participants] — Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Maintain Weight or Experience Weight Gain
Description: A patient will be defined as "success" if he/she maintains or gains weight at the end if Initial Treatment compared with baseline of study entry.
Time Frame: 4 weeks
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: BMI Trends
Time Frame: 4 weeks
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Caloric Intake
Time Frame: 4 weeks
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Weight Maintenance Over Time
Time Frame: 4 weeks
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Toxicity Profile
Description: Number of patients with grade 3+ non-hematologic adverse events using Common Toxicity Criteria for Adverse Effects (CTCAE) v.4.0
Time Frame: 4 weeks
Population: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Since only one patient was accrued, patient confidentiality prevents the reporting of this patient.
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes